CLINICAL TRIAL: NCT05341947
Title: A Phase I Trial of Activated Autologous T Cells Against Glioma Cancer Stem Cell Antigens for Patients With Recurrent Glioblastoma
Brief Title: Activated Autologous T Cells Against Glioma Cancer Stem Cell Antigens for Patients With Recurrent Glioblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Jeremy Rudnick, M.D (Other)
Collaborators: Kairos Pharma (Unknown)
Responsible Party: Sponsor-Investigator, Jeremy Rudnick, M.D, Co-Director, Neuro-Oncology, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2019-23-Rudnick-ATC
Record Dates: First submitted 2022-03-24; First posted 2022-04-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Glioblastoma
Keywords: glioma; brain tumor; glioblastoma; neurosurgery; surgical resection; Complete resection of tumor; extent of resection; maximal safe resection; neuropathology; astrocytoma; ependymoma
MeSH Terms: conditions — Glioblastoma; Glioma; Brain Neoplasms; Astrocytoma; Ependymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Activated T cells (Experimental)
  Interventions: Biological: Activated T cells

INTERVENTIONS:
Biological: Activated T cells — Activated T cells (ATC) administered intravenously at one timepoint

SUMMARY:
The purpose of this study is to examine the use of activated T cells (ATCs) to assess the safety and tolerability of autologous activated T cells, as measured by the number of Grade 3 or higher toxicities, the number of serious adverse events, and treatment-related toxicities, according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 5, to find the maximum tolerated dose. The secondary objectives include evaluating the rate of overall survival, rate of progression-free survival, health-related quality of life parameters, overall response rate, immune response, and tumor stem cell antigen expression.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent glioblastoma
* HLA-A1 and HLA-A2 positive
* Complete resection of tumor

Exclusion Criteria:

* Clinically significant pulmonary, cardiac or other systemic disease
* Presence of an acute infection requiring active treatment with antibiotics/antivirals; prophylactic administration is allowed.
* Known human immunodeficiency virus positivity or acquired immunodeficiency syndrome related illness or other serious medical condition.
* Known history of Hepatitis B or Hepatitis C
* Allergy to Dimethyl sulfoxide (DMSO)
* Allergy to gentamicin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Grade 3 or higher toxicities, number of serious adverse events, and the number of treatment-related toxicities to find the maximum tolerated dose | From start of study treatment until End of Study, an average of 2 months
  Recorded and graded according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAEs) Version 5

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of enrollment to date of death of any cause or withdrawal of consent, whichever came first. Assessed up to 3 years.
Progression-Free Survival (PFS) | From start of study treatment, until confirmation of disease progression or withdrawal of consent, whichever came first. Assessed up to 3 years.
Health-related quality of life parameters | From baseline visit to End of Study, an average of 2 months
  Measured by change in the Functional Assessment of Cancer Therapy - Brain (FACT-Br) survey score. The FACT-Br total score has a range of 0-200 and higher scores indicate better quality of life
Overall Response Rate (ORR) | From pre-study Brain MRI through study completion or withdrawal of consent, whichever came first. Assessed up to 3 years.
  Percentage of patients showing either partial response or complete response, in patients with subtotal resection, will be measured using Magnetic Resonance Imaging (MRI) and Immunotherapy Response Assessment in Neuro-Oncology (iRANO) Response Criteria
Immune Response | At Visit 1, Post-immunotherapy infusion follow-up Day 14, and Survival follow-up Month 2
  Assessed by cytotoxic T cell activity in vitro pre- vs post-infusion.
Tumor stem cell antigen expression | At Baseline visit and at time of recurrence. Assessed up to 3 years.
  Assessed by quantitative PCR for expression of CD133, housekeeping genes, and tumor associated antigens (including HER2, TRP-2, gp100, MAGE-1, IL13Rα2, AIM-2).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Rudnick, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States